CLINICAL TRIAL: NCT03370952
Title: Laparoscopy-assisted Ovarian Cystectomy: NEW APPROCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new approach (Active Comparator): Under general anaesthesia, the patient is placed in the modified dorsal lithotomy position a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).
  Aspiration of the cyst:
  Delivery of affected ovary outside the abdominal cavity:
  A transverse mini-laparotomy is done (2-3 cm) in the midline 2 cm above the symphysis pubis.
  Ovarian cystectomy:
  Re-introduction of the ovary to inside the abdominal cavity:
  Interventions: Procedure: combined laproscopic and minilaparotomy ovarian cystectomy
- Laproscopic ovarian cystectomy (Active Comparator): classic laparoscopic ovarian cystectomy
  Interventions: Procedure: laproscopy

INTERVENTIONS:
Procedure: laproscopy — laparoscopic ovarian cystectomy
  Arms: Laproscopic ovarian cystectomy
Procedure: combined laproscopic and minilaparotomy ovarian cystectomy — Under general anaesthesia, the patient is placed in the modified dorsal lithotomy position a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).
  Aspiration of the cyst:Delivery of affected ovary outside the abdominal cavity:
  Ovarian cystectomy:
  Re-introduction of the ovary to inside the abdominal cavity:
  Arms: new approach

SUMMARY:
Under general anaesthesia, the patient is placed in the modified dorsal lithotomy position a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).

Aspiration of the cyst:

Veress needle is inserted in the midline 2 cm above the symphysis pubis to aspirate the cyst under laparoscopic guidance (to guide the entry of the needle into the cyst wall & to confirm complete aspiration).

Delivery of affected ovary outside the abdominal cavity:

Classic ovarian cystectomy will be done using microsurgical techniques in which the cyst wall will be dissected gently and carefully from the healthy ovarian tissue followed by perfect haemostasis and re-fashioning of the remaining ovarian tissue using Vicryl (3-0) sutures.

Re-introduction of the ovary to inside the abdominal cavity:

The stitched ovary is pushed gently inside the abdominal cavity and the mini-laparotomy is re-covered by the rubber shield (to allow re-inflation of the abdominal cavity). The ovary is reassessed under laparoscopic guidance to ensure perfect haemostasis and normal position of the ovary. Pelvic irrigation is done if needed.

DETAILED DESCRIPTION:
Patient positioning and port placement:

Under general anaesthesia, the patient is placed in themodified dorsal lithotomy position (to ensure lax anterior abdominal wall). The patient is thenprepped and draped in the usual fashion for an abdominaland vaginal procedure. In non- virgin patients, vaginal speculum is inserted into thevagina to expose the cervix, a uterine manipulator is inserted in the cervix followed by placement of a Foley's catheter in thebladder. As regards port placement, a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).

Aspiration of the cyst:

Veress needle is inserted in the midline 2 cm above the symphysis pubis to aspirate the cyst under laparoscopic guidance (to guide the entry of the needle into the cyst wall & to confirm complete aspiration).

Delivery of affected ovary outside the abdominal cavity:

A transverse mini-laparotomy is done (2-3 cm) in the midline 2 cm above the symphysis pubis. A long shanks artery forceps is introduced inside the abdominal cavity (to grasp the affected ovary) under laparoscopic guidance. Then, the artery is pulled gently to the outside to deliver the ovary at the mini-laparotomy skin incision. Careful handling and traction is applied to avoid injury of both the ovarian tissue or/andinfundibulopelvic ligament. Following the delivery of the ovary, the abdominal incision is temporary closed using (E-shaped 10 x 10 cm) rubbershield (to avoid any soiling of abdominal cavity with blood or cystic fluid & give the chance to reinflate the abdominal cavity later on).

Ovarian cystectomy:

Classic ovarian cystectomy will be done using microsurgical techniques in which the cyst wall will be dissected gently and carefully from the healthy ovarian tissue followed by perfect haemostasis and re-fashioning of the remaining ovarian tissue using Vicryl (3-0) sutures.

Re-introduction of the ovary to inside the abdominal cavity:

The stitched ovary is pushed gently inside the abdominal cavity and the mini-laparotomy is re-covered by the rubber shield (to allow re-inflation of the abdominal cavity). The ovary is reassessed under laparoscopic guidance to ensure perfect haemostasis and normal position of the ovary. Pelvic irrigation is done if needed.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral ovarian cysts (≥ 10 cm),
* recurrent ovarian cysts
* good ovarian reserve (antimullerian hormone {AMH} > 1 ng/ml & antral follicular count {AFC} > 4)

Exclusion Criteria:

* solid ovarian masses
* patients who were unfit for surgery
* chronic diseases (e.g. cardiac disease or diabetes)
* any contraindication for laparoscopic surgery (excessive anterior abdominal wall scarring)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
recurrence of ovarian masses | 6 months after the operation
  recurrence was defined as the presence of ovarian cysts ≥2 cm in the ipsilateral ovary

SECONDARY OUTCOMES:
serum follicle stimulating hormone | 6 months after the operation
  Measurement of FSH on 2nd day of a natural cycle as a marker of ovarian reserve
Serum antimullerian hormone | 6 months after the operation
  Measurement of AMH on 2nd day of a natural cycle as a marker of ovarian reserve

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Study Director — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shaltout MF, Maged AM, Abdella R, Sediek MM, Dahab S, Elsherbini MM, Elkomy RO, Zaki SS. Laparoscopic guided minilaparotomy: a modified technique for management of benign large ovarian cysts. BMC Womens Health. 2022 Jul 4;22(1):269. doi: 10.1186/s12905-022-01853-4. PMID 35787807